CLINICAL TRIAL: NCT04294095
Title: My Baby My Move A Community Wellness Intervention
Acronym: MBMM+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 19-1366; 1R21HD097450-01A1 (NIH)
Record Dates: First submitted 2020-01-23; First posted 2020-03-03 (Actual); Results first posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Gestational Weight Gain
MeSH Terms: conditions — Gestational Weight Gain

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial (control and intervention)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): During the first four weeks of the MBMM+ program, participants will receive electronic informational handouts covering topics on weight management as well as the benefits and safety concerns related to prenatal physical activity. Starting week 5 of the 12-week intervention, participants will attend two in-person, group physical activity sessions per week with each session lasting approximately 60 minutes and will be held at a local community center located close to the recruitment clinics. Sessions will be held on weekday evenings and weekend mornings as these times were preferred by pregnant women. Each session will include both didactic and experiential components to increase knowledge and skill building.
  Interventions: Other: My Baby My Move +
- Control (Active Comparator): Electronic materials related to various prenatal topics including preparation for birth, birthing options, and responsive parenting will be distributed twice a week for the first 4-weeks of the program. Starting week 5 of the 12-week intervention, participants will attend two in-person, group sessions per week with each session lasting approximately 60 minutes and will be held at a local community center located close to the recruitment clinics.
  Interventions: Other: Control

INTERVENTIONS:
Other: My Baby My Move + — This is a community-based, peer-led 12-week wellness intervention to decrease excessive gestational weight gain.
  Arms: Intervention
Other: Control — This is a 12-week basic prenatal education class.
  Arms: Control

SUMMARY:
My Baby, My Move+ (2019-2021) is a peer-led wellness intervention which aims to reduce excessive gestational weight gain (EGWG) by targeting prenatal physical activity, mood, and sleep quality. Up to 50% of pregnant women in the U.S. gain weight in excess of the Institute of Medicine guidelines. EGWG leads to poor maternal and child outcomes. It also sets the stage for long-term overweight/obesity for both mother and child. The MBMM+ intervention is an example of a theoretically-based prenatal physical activity intervention that targets these outcomes.

Up to 100 pregnant women (50 intervention arm, 50 control arm) will be recruited from the University of Colorado Clinics. Women in the intervention arm will participate in the 12-week MBMM+ intervention. Leiferman and her team propose to develop and test the feasibility and sustainability of the MBMM+ intervention to instill good healthy habits (e.g., prenatal physical activity, good sleep hygiene, stress management) during and beyond pregnancy. Findings from this study will be used to inform a future, large randomized trial.

DETAILED DESCRIPTION:
Intervention Group:

The MBMM+ intervention is designed to promote the engagement in physical activity and takes into account barriers among pregnant women cited in our formative work such as lack of knowledge and skills, body changes and discomfort, feeling limited, and lack of social support. Uniquely, the MBMM+ program also targets sleep hygiene and mood to further support regular physical activity engagement. Over the years of working with pregnant women, we have observed that once women notice how their regular physical activity helps their mood and sleep patterns they are often more likely to continue engaging in regular physical activity. During the first four weeks of the MBMM+ program, participants will receive electronic informational handouts covering topics on weight management (content will be based in part on Co-I Downs' Healthy Mom Zone intervention such as informing on benefits and guidelines of healthy GWG, tips on healthy eating, energy balance, and sleep quality) as well as the benefits and safety concerns related to prenatal physical activity. Starting week 5 of the 12-week intervention, participants will attend two in-person, group physical activity sessions per week with each session lasting approximately 60 minutes and will be held at a local community center located close to the recruitment clinics. Sessions will be held on weekday evenings and weekend mornings as these times were preferred by pregnant women. Given that pregnant women often express a lack of knowledge about safe physical activities during pregnancy, preventing them from engaging in physical activity, each session will include both didactic and experiential components to increase knowledge and skill building. Sessions will begin with a didactic component covering overcoming barriers to physical activity, goal setting, self-monitoring, problem solving, topics related to mood (stress management, family/work balance, wellness wheel), sleep hygiene (setting routines, avoiding stimulants, environmental supports), and additional physical activity topics (e.g., managing physical activity in postpartum, overcoming relapses). Participants will be given educational materials in print and electronic form based on their preferences. The experiential component (i.e., physical activity) will be 30 minutes in duration and involve primarily walking, at a moderate intensity, based on national recommendations coupled with yoga. Our formative work suggests that mothers prefer walking and find it more enjoyable in the form of groups. We have chosen to also include yoga to provide options for ways to be active that also positively impact sleep and mood and pregnant women report desiring prenatal yoga. All walking sessions will be facilitated by the peer leaders. The yoga sessions will be taught by an experienced prenatal yoga instructor residing in Denver, CO.

Each session will have 3-4 peer leaders to help facilitate and model the physical activity component (i.e., will accompany women during their walking and yoga sessions to provide support and ensure safety (e.g., correct postures during yoga, monitoring exercise intensity and symptoms during walking sessions). Our MBMM formative work and expertise in community-based physical activity interventions suggests participants prefer peer group leaders because they foster a sense of community and social support within the group setting. Peer leaders will be compensated for their time working with the MBMM+ program and will be peer mothers from the community who are recent mothers (< two years postpartum) who successfully engaged in regular physical activity during a previous pregnancy. Peer leaders will be identified by our research team, recreation center directors, and health care provider partners. At the end of every session, participants will check in with an assigned peer leader to discuss in small groups their weekly logs. Peer leaders will note the discussions that occurred amongst the participants in their group, describe barriers that were identified, problem-solving strategies that were suggested and used, and future goals/recommended action steps. This group work will help participants to learn ways to fit physical activity into their lifestyle and overcome barriers by receiving feedback from their peer leader and other group members. It will also ensure that the intervention is conducted and received in the way intended as the peer leaders and program manager/PI will review these small group progress notes each week and monitor intervention delivery.

Peer leader training and fidelity: Weekly, the research team (PI/program manager) will have phone calls and/or in-person meetings with the group peer leaders to debrief and address any issues that may arise. The program manager and/or PI will be on-site for all sessions to ensure quality control of intervention delivery and data collection efforts by peer leaders. The PI will conduct a training session before the onset of the intervention with the peer group leaders to cover topics including how to engage in safe and effective physical activity during pregnancy, an overview of behavioral change theory and the behavioral skills that the intervention is targeting, ways to garner social support and leadership skills. The PI has been extensively trained by the Cooper Institute in Prenatal-Postnatal Physical Activity. The yoga instructor will have been extensively trained in prenatal yoga.

Control Group:

Women randomized to the control group will complete a similarly structured 12-week program; electronic materials related to various prenatal topics including preparation for birth, birthing options, and responsive parenting will be distributed twice a week for the first 4-weeks of the program. Starting week 5 of the 12-week intervention, participants will attend two in-person, group sessions per week with each session lasting approximately 60 minutes and will be held at a local community center located close to the recruitment clinics. Sessions will be held on weekday evenings and weekend mornings as these times were preferred by pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* pregnant (6-10 weeks) women
* aged 18-46 years
* reside in Denver, CO
* currently engaging in less than 120 minutes of moderate-intensity exercise per week
* have medical clearance to exercise during pregnancy.

Exclusion Criteria:

-having conditions that preclude exercise (i.e. HCP has restricted patient from engaging in exercise according to AGOG's absolute contraindications to exercise (e.g. haemodynamically significant heart disease, restrictive lung disease, incompetent cervix/cerclage, persistent second or third trimester bleeding, placenta previa after 26 weeks gestation, premature labor during the current pregnancy, ruptured membranes, and pregnancy induced hypertension)

Ages: 18 Years to 46 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant Women
Enrollment: 68 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jenn Leiferman, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other researchers

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 68 participants were consented - 18 dropped out prior to randomization due to physician request, no longer interested A total of 50 participants were randomized of which 49 completed all assessments.
Groups:
- Intervention: During the first four weeks of the MBMM+ program, participants will receive electronic informational handouts covering topics on weight management as well as the benefits and safety concerns related to prenatal physical activity. Starting week 5 of the 12-week intervention, participants will attend two in-person, group physical activity sessions per week with each session lasting approximately 60 minutes and will be held at a local community center located close to the recruitment clinics. Sessions will be held on weekday evenings and weekend mornings as these times were preferred by pregnant women. Each session will include both didactic and experiential components to increase knowledge and skill building. Please note that in-person sessions were moved to online platform for the entire trial due to covid.
  My Baby My Move +: This is a community-based, peer-led 12-week wellness intervention to decrease excessive gestational weight gain.
- Control: Electronic materials related to various prenatal topics including preparation for birth, birthing options, and responsive parenting will be distributed twice a week for the first 4-weeks of the program. Starting week 5 of the 12-week intervention, participants will attend two in-person, group sessions per week with each session lasting approximately 60 minutes and will be held at a local community center located close to the recruitment clinics.
  Control: This is a 12-week basic prenatal education class. Please note that in-person sessions were moved to online platform for the entire trial due to covid.
Period: Overall Study
Arm/Group | Intervention | Control
Started | 26 | 24
Completed | 25 | 24
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 25 | 24 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.1 (4.87) | 31.5 (4.3) | 31.8 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 24 | 49
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 7 | 4 | 11
  nonHispanic | 18 | 20 | 38
Region of Enrollment [Number; unit: participants]
  United States | 25 | 24 | 49
Weight [Count of Participants; unit: Participants]
  Underweight | 2 | 2 | 4
  Normal Weight | 11 | 15 | 26
  Overweight | 8 | 3 | 11
  Obese | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Weight
Description: Average weight
Time Frame: 12 week post-baseline
Population: Average Weight of pregnant women for intervention versus control at 12 weeks post-baseline
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Intervention | Control
Number analyzed (Participants) | 25 | 24
pounds | 162.9 (29.9) | 162.3 (37.6)

2. Secondary Outcome: Depression
Description: Edinburgh Postnatal Depression Scale (EPDS); scale: 1-30 with higher score indicating higher depression
Time Frame: 12 weeks post-baseline
Population: Depression scores at 12 wks post baseline for intervention vs control
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 25 | 24
units on a scale | 8.1 (5.4) | 6.3 (4.4)

3. Secondary Outcome: Anxiety
Description: General Anxiety Disorder- 7 scale (GAD-7); 1-7 scale with higher score indicating higher anxiety
Time Frame: 12 weeks post baseline
Population: 12 wk post-baseline anxiety scores for intervention and control
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 25 | 24
units on a scale | 4.7 (3.1) | 3.7 (3.2)

4. Secondary Outcome: Physical Activity
Description: The Godin-Shephard Leisure-Time Physical Activity Questionnaire (LTEQ) assesses when someone engages in mild, moderate, and vigorous exercise for more than 15 minutes within one week. The leisure activity score is calculated using the following formula: leisure activity score = (9 x strenuous activity per week) + (5 x moderate activity per week) + (3 x light activity per week). Strenuous exercise is defined as heart beating rapidly, moderate exercise is defined as not exhausting, and light activity is described as minimal effort. Scores of 14 or less indicate insufficiently active/sedentary, scores of 14-23 indicate moderately active, and scores of more than 24 indicate active.
Time Frame: 12 weeks Post-baseline
Population: 12 weeks post-baseline assessment of physical activity for intervention and control.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 25 | 24
units on a scale | 48.0 (17.8) | 35.9 (9.11)

ADVERSE EVENTS:
Time Frame: 16 months
Description: serious adverse event - miscarriage.
Groups:
- Intervention: During the first four weeks of the MBMM+ program, participants will receive electronic informational handouts covering topics on weight management as well as the benefits and safety concerns related to prenatal physical activity. Starting week 5 of the 12-week intervention, participants will attend two in-person, group physical activity sessions per week with each session lasting approximately 60 minutes and will be held at a local community center located close to the recruitment clinics. Sessions will be held on weekday evenings and weekend mornings as these times were preferred by pregnant women. Each session will include both didactic and experiential components to increase knowledge and skill building. Please note that all in-person sessions were moved to an online platform due to Covid.
  My Baby My Move +: This is a community-based, peer-led 12-week wellness intervention to decrease excessive gestational weight gain.
- Control: Electronic materials related to various prenatal topics including preparation for birth, birthing options, and responsive parenting will be distributed twice a week for the first 4-weeks of the program. Starting week 5 of the 12-week intervention, participants will attend two in-person, group sessions per week with each session lasting approximately 60 minutes and will be held at a local community center located close to the recruitment clinics. Please note that all in-person sessions were moved to an online platform due to Covid.
  Control: This is a 12-week basic prenatal education class.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/24
Serious Adverse Events (participants affected / at risk) | 1/25 | 0/24
Other Adverse Events (participants affected / at risk) | 0/26 | 0/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=25) | Control (N=24)
miscarriage (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) — Miscarriage

LIMITATIONS AND CAVEATS:
The trial was limited due to the onset of the Covid pandemic and the inability to have direct contact with participants. The entire trial had to pivot from an in-person data collection and intervention delivery system to an online platform and limited objective data collection. Due to the special population of pregnant women and the associated high-risk of covid, we had challenges recruiting women as well as obtaining medical clearance forms from overburdened health care providers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-06): https://cdn.clinicaltrials.gov/large-docs/95/NCT04294095/Prot_SAP_001.pdf
  • Informed Consent Form (2021-02-25): https://cdn.clinicaltrials.gov/large-docs/95/NCT04294095/ICF_000.pdf